CLINICAL TRIAL: NCT00575120
Title: Assessment of Endothelial Function Using Blood Oxygen Level-Dependent MRI (BOLD-MRI)
Brief Title: Endothelial Function Assessed With BOLD-MRI
Acronym: EFBOLD-MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Oliver Strohm, Adunct Research Associate Professor, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: E-21003; Protocol #21003
Record Dates: First submitted 2007-12-10; First posted 2007-12-18 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: Endothelial Function
Keywords: Endothelial Function, MRI, Vascular Biology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (No Intervention): Endothelial Function of forearm assessed by FMD, PAT, BOLD-MRI before 15 min. ischemia reperfusion of forearm
- B (Active Comparator): Endothelial Function of forearm assessed by FMD, PAT, BOLD-MRI after 15 min. ischemia reperfusion
  Interventions: Other: ischemia reperfusion

INTERVENTIONS:
Other: ischemia reperfusion — reperfusion after a 15 min. lasting cuff induced arm ischemia
  Other Names: CMR imaging study
  Arms: B

SUMMARY:
The purpose of this study is to assess the applicability of a new SSFP-based BOLD sensitive MRI sequence in evaluating endothelial function. Endothelial function will be tested in a setting of reactive hyperemia in the forearm. In a setting of ischemia-reperfusion, the effect of transient endothelial function impairment will be tested. Comparison with endothelial function assessment by brachial ultrasound (FMD) and finger tip plethysmography (PAT) will be incorporated.

Hypothesis: BOLD-MRI is a feasible tool to assess endothelial function in the human forearm during reactive hyperemia. There is significant correlation to established flow-mediated dilation (FMD).

DETAILED DESCRIPTION:
This is a single center study on healthy volunteers. The subjects will be seen by the study coordinator in the SCMRC to obtain written informed consent and to assess the co-variable data (vitals, medication, history, contraindications for MRI). The study nurse will schedule two visits for endothelial function assessment that are at least one but not more than three weeks apart. Both visits are to be at the same time of day. The initial volunteer will be assigned an endothelial function assessment with MRI first followed by FMD in the endothelial function lab. Subsequent volunteers will alternate assignment to FMD or MRI first to rule out pre-conditioning effects. Simultaneous to FMD assessment, plethysmographic pulse volume will be evaluated with finger probes on the index finger of each hand. Subjects will be studied in a temperature-controlled room with minimal background distraction and in a fasting state for the previous 4 hours. Subjects will also refrain from ingesting caffeine or nicotine in these preceding 4 hours. Each study day volunteers will undergo two endothelial function assessments. The first baseline assessment takes place after a 10 minute accommodation period. The volunteer is then subjected to a 15 minute upper arm tourniquet. The second assessment takes place 15 minutes after the release of the tourniquet. This so called 'ischemia reperfusion' is known to markedly impair endothelial function for approximately one hour without affecting the early bloodflow responses to reactive hyperemia. This effect is reversible and will help to determine the actual endothelial component of measured BOLD signal changes.

One day: 2 CMR studies without contrast agent to assess endothelial function during reactive hyperemia. Each will last 15 minutes. A 15 minutes upper arm occlusion with a pressure cuff in between the 2 measurements will be applied.

Another day: 2 FMD studies with ultrasound to assess endothelial function during reactive hyperemia. Each will take 15 minutes. Simultaneously a PAT hyperemic index will be measured. A 15 minutes upper arm occlusion with a pressure cuff in between the 2 measurements will be applied.

Blood work (fasting glucose, creatinine, lipids, hsCRP), performed by Calgary Labs Services (CLS).

The effect of the reperfusion ischemia will be tested by individually comparing the BOLD signal change (BC) at baseline with BC after reperfusion ischemia. Since these are paired, related data a Wilcoxon rank sum test will be performed and a p value < 0.05 will be regarded as significant. The same will be done for the FMD and PAT index before and after reperfusion ischemia.

FMD as the most accepted technique and will be considered as gold standard and a linear regression analysis of FMD with MBC and TBC will be performed. r2-value will be calculated and a value of > 0.25 will be considered as reasonable of > 0.5 as good correlation. If the correlation does not appear linear a Spearman's correlation test will be done.

The correlations between PAT index and FMD and PAT index and TBC will also be assessed with linear regression analysis.

ELIGIBILITY:
Inclusion criteria

* Informed written consent
* male gender
* age > 18 years
* fasting for 4 hours prior to the study and especially no coffee

Exclusion criteria

* Contraindications for MRI
* female gender
* known cardiovascular disease including: CHD, congestive heart failure, peripheral vascular disease
* known cardiovascular risk factors : smoking, diabetes mellitus, hypertension, hyperlipidemia
* Current vasoactive medication : Beta-blockers, Ca-Antagonists, ACE-Inhibitors, ARB, Phosphodiesterase inhibitors
* concomitant serious medical condition
* unreliability as a volunteer or inability or unwillingness to complete the study and the second day of examination

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
BOLD-MRI signal-intensity | 75 min

SECONDARY OUTCOMES:
FMD PAT | 75 min

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Friedrich, MD, Principal Investigator — University of Calgary
Locations (1):
- Stephenson CMR Centre at Foothills Medical Centre, University of Calgary, Calgary, Alberta, Canada